CLINICAL TRIAL: NCT00644735
Title: Multicenter, Randomized, Double-Blind, Double-Dummy, Parallel-Group Comparison of the Remission Rates of Once Daily Treatment With Esomeprazole 20mg and Lansoprazole 15mg for 6 Months in Patients Whose EE Has Been Healed.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, Astra Zeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 325; D9612L00048
Record Dates: First submitted 2008-03-18; First posted 2008-03-27 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Erosive Esophagitis
Keywords: Erosive Esophagitis; Nexium; Esomeprazole; Lansoprazole; Heartburn
MeSH Terms: conditions — Heartburn | interventions — Esomeprazole; Lansoprazole

ARMS (2):
- 1 (Experimental): Nexium
  Interventions: Drug: Esomeprazole
- 2 (Active Comparator): Prevacid
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Esomeprazole
  Other Names: Nexium
  Arms: 1
Drug: Lansoprazole
  Other Names: Prevacid
  Arms: 2

SUMMARY:
A study to look at the rates of remission (non re-appearance of erosive esomeprazole) when treated with esomeprazole or lansoprazole; in patients in with erosive esomeprazole (EE) that is in remission (i.e. previously healed EE).

ELIGIBILITY:
Inclusion Criteria:

* Episodes of heartburn (described as a burning feeling rising from the stomach or lower part of the chest up towards the neck) for 2 days or more during the last 7 days prior to baseline
* Confirmed diagnosis of Erosive Esophagus, patients must undergo an endoscopy before entering the study.

Exclusion Criteria:

* Any signs of gastrointestinal bleeding at the time of the starting the study.
* Any previous gastric or esophageal surgery.
* Various gastrointestinal diseases as listed in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2002-12; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
To compare rates of remission (non re-appearance of erosive esomeprazole) when treated with esomeprazole or lansoprazole; in patients in with erosive esomeprazole (EE) that is in remission (i.e. previously healed EE). | Symptoms will be assessed by the investigator at each visit and the patients will undergo an endoscopy at Months 3 and 6

SECONDARY OUTCOMES:
To compare endoscopic remission rates through 6 months of treatment with E20 and L15, after initial healing of EE. | Symptoms will be assessed by the investigator at each visit and the patients will undergo an endoscopy at Months 3 and 6
The assessment of symptoms in the two treatment groups after 1, 3 and 6 months. | patients will undergo an endoscopy at Months 3 and 6
To assess the safety and tolerability of up to 6 months of treatment with E20 and L15 after initial healing of EE. | Symptoms will be assessed by the investigator at each visit and the patients will undergo an endoscopy at Months 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca